CLINICAL TRIAL: NCT02692443
Title: Single Ventricle Reconstruction III: Brain Connectome and Neurodevelopmental Outcomes
Brief Title: SVR III: Brain Connectome and Neurodevelopmental Outcomes
Acronym: SVRIII
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Boston Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Emory University (Other); Medical College of Wisconsin (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Ashok Panigrahy, Associate Professor of Radiology, University of Pittsburgh
Other Study IDs: R01HL128818 (NIH)
Record Dates: First submitted 2015-09-24; First posted 2016-02-26 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Magnetic Brain Resonance; CHD; MRI; Neurodevelopmental
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SVR Survivors: Through the SVR and SVR II studies vital status has been followed annually for the entire SVR cohort. As of June 2014 352 subjects are alive, 18 of whom have undergone cardiac transplantation, and 18 have undergone biventricular conversion leaving 334 transplant-free survivors with single ventricle physiology. Each patient enrolled to this ancillary study from the parent SVR study will be asked to undergo Magnetic Resonance Imaging (Brain MRI without Contrast) in addition to the already scheduled parent study follow-up procedures.
  Interventions: Device: Magnetic Resonance Imaging; Behavioral: Neurodevelopmental Testing
- Healthy Controls: In addition to the SVR survivors, investigators plan to enroll 100 age- and gender-matched healthy controls. Healthy controls enrolled for participation in this ancillary study will be asked to undergo Magnetic Resonance Imaging (Brain MRI without Contrast) in addition to completing the Neurodevelopmental Testing Battery that is already part of the parent SVR study and completed by SVR Survivors as part of their SVR follow-up appointments.
  Interventions: Device: Magnetic Resonance Imaging; Behavioral: Neurodevelopmental Testing

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Brain MRI without Contrast
Behavioral: Neurodevelopmental Testing — Validated battery of neurodevelopmental and psychological tests.

SUMMARY:
Patients with hypoplastic left heart syndrome and other single right ventricle lesions who have undergone the Fontan procedure have a high risk of neurodevelopmental disorders that affect quality of life and adulthood employment. This study will leverage the ongoing National Heart, Lung, and Blood Institute (NHLBI)-funded Single Ventricle Reconstruction Study by using innovative graph measures of brain connectivity to elucidate how alterations of the "connectome" in children with critical congenital heart disease are associated with developmental disabilities and their associated clinical risk factors. Improved understanding of these interrelationships may facilitate development of targeted interventions to improve outcome in the soaring population of adult Fontan survivors.

DETAILED DESCRIPTION:
With dramatic improvement in survival of patients with hypoplastic left heart syndrome and related forms of single right ventricle undergoing staged palliation to the Fontan operation, a high prevalence of neurodevelopment abnormalities has been exposed. The NHLBI-funded Pediatric Heart Network (PHN) Single Ventricle Reconstruction (SVR) III study, "Long-term Outcomes of Children with Hypoplastic Left Heart Syndrome (HLHS) and the Impact of Norwood Shunt Type," is a prospective follow-up study of an existing cohort of children with HLHS and other single RV anomalies who were enrolled in early infancy in a randomized clinical trial of the modified Blalock-Taussig shunt (MBTS) versus right ventricular to pulmonary artery shunt (RVPAS). The parent SVR III study seeks to determine if the shunt assignment at the time of the Norwood operation is associated with cardiac function, transplant-free survival, exercise function, and neurodevelopmental outcomes. The investigators here propose a neuroimaging ancillary study to the parent SVRIII study that leverages the neurodevelopmental follow-up of the SVR cohort at age 11 years. The investigators will combine state-of-the-art brain imaging techniques [Resting-Blood Oxygenation Level Dependent (BOLD) and Diffusion Tensor Imaging] in 140 SVR III patients and 100 referent subjects with innovative brain connectome or "graph" analyses to determine if brain connectivity graph measurements will provide novel neuroimaging biomarkers for neurodevelopmental disabilities and improve the investigators' understanding of their inciting mechanisms in the SVR survivors. The investigators' specific aims are: Specific Aim (SA) #1: To characterize the global brain network topology of the SVR III cohort; SA #2: To determine which neurocognitive and behavioral outcomes predict global brain network topology in the SVR III cohort. SA #3: To determine which patient factors (e.g., birth weight, gestational age, maternal education) and medical factors (e.g., intraoperative conduct during Norwood procedure, hemodynamic complications, types and number of interventions, and measures of global morbidity) predict global brain network topology in the SVRIII cohort. SA #4: To precisely characterize the specific relationships between global brain network topology, specific patient/medical factors, and adverse neurocognitive/behavioral outcomes in the SVRIII cohort. The investigators will use linear regression and mediation statistical methods to analyze associations of MRI graph measures with SVRIII neurodevelopmental measures and surgical/non-surgical clinical independent risk factors. Upon successful completion, these studies will elucidate the nature and basis of neurodevelopmental disability in single ventricle patients following Fontan palliation. This research will also contribute a novel and robust set of clinical/research tools in the form of neuroimaging biomarkers that can be used to help classify and predict outcomes in complex congenital heart disease (CHD).

ELIGIBILITY:
Inclusion Criteria:

* SVR Survivor:
* All SVR study cohort members will be contacted to assess for vital status
* Transplant free survivors will be approached to participate in the in-person assessment
* Healthy Controls: Males and females aged 10 - 12 at the time of enrollment and whose parent or legal guardian can provide consent for participation will be recruited for participation in this study. Study participants will also be asked to provide assent for participation in this study.

Exclusion Criteria:

* SVR Survivors: The investigators will exclude patients who have undergone cardiac transplantation or biventricular conversion from all outcomes other than vital status.
* Those patients with a contraindication to MRI (i.e., claustrophobia; metal screen failure; inability to lie still) will not be enrolled for participation in this study.
* Healthy Controls: Potential participants will be excluded for any of the following reasons:

  1. disorders that would prevent successful completion of the planned study testing (e.g., pacemaker, metal implants; claustrophobia; inability to lie still)
  2. other forms of congenital heart disease requiring surgical correction
  3. Lack of reading fluency in English by primary caregiver in English

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: SVR Survivor - male and female - 10 to 12 years of age
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2015-08; Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
MRI and neurodevelopmental outcomes in CHD patients as compared to their healthy counterparts | Through study completion, an average of 4 years
  To precisely characterize the specific relationships between global brain network topology, specific patient/medical factors, and adverse neurocognitive/behavioral outcomes in the SVRIII cohort.

IPD SHARING:
Plan to Share IPD: Yes
Data will be supplied in the required, standard de-identified format and made available without cost to researchers or analysts. Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes.
Supporting Information: Study Protocol, SAP
Time Frame: After all study subjects have completed participation and analysis have been completed.
Access Criteria: Data will be shared through secure website with interested research and accessible only by username and password provided by PI research team.

REFERENCES:
- [Derived] Schmithorst V, Ceschin R, Lee V, Wallace J, Sahel A, Chenevert T, Parmar H, Berman JI, Vossough A, Qiu D, Kadom N, Grant PE, Gagoski B, LaViolette P, Maheshwari M, Sleeper LA, Bellinger D, Ilardi D, O'Neil S, Miller TA, Detterich J, Hill KD, Atz AM, Richmond M, Cnota J, Mahle WT, Ghanayem N, Gaynor W, Goldberg CS, Newburger JW, Panigrahy A. Single Ventricle Reconstruction III: Brain Connectome and Neurodevelopmental Outcomes: Design, Recruitment, and Technical Challenges of a Multicenter, Observational Neuroimaging Study. medRxiv [Preprint]. 2023 Apr 17:2023.04.12.23288433. doi: 10.1101/2023.04.12.23288433. PMID 37131744